CLINICAL TRIAL: NCT03725514
Title: Short Term Success of Inflamed Mature Single Rooted Teeth With Symptomatic Apical Periodontitis Following Single Visit Regenerative Treatment Protocols (Randomized Clinical Trial)
Brief Title: Evaluation of the Survival of Inflamed Mature Single Rooted Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Omar Fahim, Assistant Lecturer of Endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO28
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Regeneration
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sealed Opaque Envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Active Comparator): Conventional blood clot technique
  Interventions: Procedure: Conventional
- PRF (Experimental): Platelet Rich Fibrin Technique
  Interventions: Procedure: PRF

INTERVENTIONS:
Procedure: Conventional — Conventional Blood Clot Technique
  Arms: conventional
Procedure: PRF — Platelet Rich Fibrin Technique
  Arms: PRF

SUMMARY:
The majority of articles present in literature concerning the enrollment of tissue engineering in the field of root canal treatment is concerned with the treatment of affected teeth with immature apex, after proper systematic search online, only 4 articles where found that are dealing with the treatment of teeth with mature apex. These 4 studies are case reports. None of these studies has been a randomized clinical trial, the gold standard of interventional trials resulting in the highest level of evidence that contributes effectively in the clinical decision-making process as to the best intervention for the patient's condition providing the most effective clinical outcomes for the satisfaction of the patient. Since that the triad of regenerative endodontics are the key of success of any attempt to regenerate pulp, 2 different maneuvers shall be done in this study.

DETAILED DESCRIPTION:
Preservation of the natural dentition had always been a primary objective in endodontic practice. When the pulp is diseased or requires removal for restorative reasons, it is replaced with an artificial filling material during conventional root canal treatment. Root canal treatment has lots of drawbacks, starting with different iatrogenic errors during endodontic procedures, weakening of remaining tooth structure which might affect the tooth survival. Also Root canal treated teeth require the placement of a post and core, which itself is doubtful whether it increases fracture resistance of the tooth or it weakens it. The most important drawback is that the survival of affected pulp is hindered by the conventional root canal treatment. Thus a new treatment approach was introduced utilizing the body ability to regenerate, called Pulp Regeneration. Regeneration was first introduced in the dental field as a solution for immature apex treatment, due to difficulties encountered during its conventional root canal treatment. Here the Pulp regeneration shall be used on vital mature teeth to increase the survival rate of the affected teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic diseases.
* Non-pregnant females
* Single canalled teeth.
* Patients having vital, mature, single rooted teeth, clinical evidence of pulpitis and apical periodontitis.
* Positive patient/Guardian compliance for participation in the study.

Exclusion Criteria:

* Any known sensitivity or adverse reactions to medicaments or pharmaceuticals necessary to complete the trial.
* Non-restorable coronal portion of teeth involved in the trial.
* Non Vital teeth
* Immature teeth
* Traumatized teeth
* Radiographic evidence of external or internal root resorption.
* Single Rooted teeth with multiple canals.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of tooth Sensitivity | 1, 3, 6, 9, 12 Months
  Electric Pulp Tester

SECONDARY OUTCOMES:
Survival | 1, 3, 6, 9, 12 Months
  Clinical examination of tooth integrity
Clinical Success | 1, 3, 6, 9, 12 Months
  Clinical examination the signs & symptoms is present or absent
Pericapical Status | 6, 9, 12 Months
  CBCT assessment in Hounsfield unit
Periapical Status | 1, 3, 6, 9, 12 Months
  Digital Periapical Radiograph in pixels

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be made available
Supporting Information: Study Protocol, ICF
Time Frame: It will be available after finishing the study
Access Criteria: It will be uploaded on a folder on google drive to be accessed through this link URL: https://drive.google.com/open? id=1rZXDbSgsneWDO4xGz8KGkklEHHw2YYIX
URL: https://drive.google.com/open?id=1rZXDbSgsneWDO4xGz8KGkklEHHw2YYIX

REFERENCES:
- [Background] Araujo PRS, Silva LB, Neto APDS, Almeida de Arruda JA, Alvares PR, Sobral APV, Junior SA, Leao JC, Braz da Silva R, Sampaio GC. Pulp Revascularization: A Literature Review. Open Dent J. 2017 Jan 31;10:48-56. doi: 10.2174/1874210601711010048. eCollection 2017. PMID 28567136